CLINICAL TRIAL: NCT04042935
Title: Alpha Lipoic Acid to Decrease Treatment Related Pain and Side Effects During Concurrent Chemoradiation in HNSCC
Brief Title: Alpha Lipoic Acid to Decrease Pain and Side Effects in Concurrent Treatment of HNSCC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Cancer League of Colorado (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-1081.cc
Record Dates: First submitted 2019-07-26; First posted 2019-08-02 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: HNSCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Thioctic Acid

STUDY DESIGN:
Intervention Model Description: 3+3 Dose Escalation: Dose Level -2: ALA 300 mg daily Dose Level -1: ALA 600 mg daily Dose Level 1: ALA 600 mg BID Dose Level 2: ALA 600 mg TID
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Alpha Lipoic Acid (ALA) during chemoradiation (Experimental): Stage II-IVB HNSCC patients receiving concurrent systemic therapy and radiation as standard of care will receive ALA before, during, and after treatment. The drug will have dose escalation in a 3+3 design. The first group of 3 patients will receive 600 mg twice a day. If there are no DLTs, the next 3 patients will receive the highest dose of 600 mg three times a day. If one or more patients develop a DLT at any of the dosing levels, the group will either be expanded or dropped to a lower dose level.
  Interventions: Drug: Alpha Lipoic Acid

INTERVENTIONS:
Drug: Alpha Lipoic Acid — Stage II-IVB HNSCC patients receiving concurrent systemic therapy and radiation in the definitive, adjuvant, or palliative setting will receive ALA according to their prescribed dose level. ALA will be taken orally or per feeding tube. It will start 1 week prior to the start of CRT, continue on through CRT, and then continue for 2 weeks after the completion of CRT. Patients will be given dosing diaries to document date and time of each drug administration as well as any missed doses. They will also have weekly visits to report AEs and concurrent medications, have a history and physical exam, report VAS pain scores and OMAS scores, and fill FACT-HN surveys.

SUMMARY:
This is a phase I, single-center, non-randomized, 3+3 dose-escalation study of alpha lipoic acid given during chemotherapy-radiation in HNSCC patients with non-metastatic disease.

DETAILED DESCRIPTION:
The study will be completed when the MTD and RP2D are determined. This will be either when 2 or more patients have a DLT at a particular dose level, or when 6 patients have completed treatment at the highest dose level (600 mg TID). The final 3 patients enrolled at the highest tolerated dose will also complete PK studies.

ELIGIBILITY:
Inclusion Criteria:

1. Provision to sign and date the consent form.
2. Stated willingness to comply with all study procedures and be available for the duration of the study.
3. Be a male or female aged 18-100.
4. Histologically or cytologically confirmed stage II-IVB HNSCC of the oral cavity, hypopharynx, oropharynx, larynx, or nasopharynx.
5. Ability to take medication orally or per feeding tube and be willing to adhere to the medication regimen.
6. Patients who are deemed appropriate for definitive, adjuvant, or palliative radiation with total planned dose > 30 Gy.
7. Patients who are deemed appropriate for concurrent systemic therapy with radiation including cisplatin (100 mg/m2 triweekly or 30-40 mg/m2 weekly), carboplatin (AUC 1-2 weekly) +/- paclitaxel (30 mg/m2 weekly) or cetuximab (400 mg/m2 loading followed by 250 mg/m2 weekly.

   a. The final 3 patients in the dose expansion group undergoing the PK/PD study must be deemed appropriate for cisplatin.
8. For females of reproductive potential: use of highly effective contraception including hormonal contraceptives, intrauterine devices (IUD), vasectomy, tubal ligation, and double barrier methods (combination of male condom, female condom, cervical cap, diaphragm, contraceptive sponge).
9. For males of reproductive potential: use of condoms.
10. ECOG performance status ≤ 2.

Exclusion Criteria:

1. Participation in another clinical study with an investigational product during the last 30 days.
2. Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study, a clinical study not involving pharmaceutical or radiation techniques, or during the follow-up period of an interventional study.
3. Women who are pregnant or lactating. Patients of reproductive potential must have a negative serum or urine pregnancy test within 72 hours of start of study drug.
4. Patients who are currently taking gabapentin, pregabalin, amitriptyline, nortriptyline, or duloxetine.
5. Known allergy or hyposensitivity to alpha lipoic acid.
6. Judgement by the investigator that the patient is unsuitable to participate in the study and the patient in unlikely to comply with study procedures, restrictions, and requirements.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2021-09-24 (Actual)

PRIMARY OUTCOMES:
MTD and RP2D of ALA during chemoradiotherapy for HNSCC patients | 18 months
  The maximum tolerated dose will be the highest dose in the planned schema that is given without evidence of SAEs.
  The RP2D will incorporate the MTD and PKs to determine the dose that is best tolerated as well as has the concentration necessary to be effective according to historical studies.

SECONDARY OUTCOMES:
Safety of ALA by following adverse events (AEs) | up to 18 months
  Adverse events will be documented to determine the primary endpoints as well as to categorize potential side effects that can be attributed to ALA. CTCAE version 5.0 will be used to categorize the AEs
Maximum plasma concentration of ALA at the MTD with chemoradiotherapy | At start of ALA, Day 1, and Day 15, for 3 dose expansion PK patients
  Maximum plasma concentration will be evaluated on the 3 patients in the dose expansion group at the MTD. This will be studied when given with cisplatin for standardization to ensure concentration is similar to when ALA is given alone.
Change in Oral Mucositis Assessment Scale (OMAS) from baseline | From start of treatment to post-treatment surveillance scans, up to 6 months
  OMAS scores will give preliminary measures on efficacy of drug to control pain and improve quality of life which will be the primary focus in future studies. Total scores will be collected from 0 (no mucositis) to 45 (worse mucositis). Average OMAS and change from baseline to worst score will be evaluated.
Change in Visual Assessment Score (VAS) for pain from baseline | From start of treatment to post-treatment surveillance scans, up to 6 months
  VAS for pain will give preliminary measures on efficacy of drug to control pain which will be the primary focus in future studies. The VAS score is from 0-10 with 0 being no pain and 10 being the worse possible pain. Average VAS and change from baseline to worst score will be evaluated.
Change in quality of life measures using the Functional Assessment of Cancer Therapy - Head & Neck (FACT-HN) during chemoradiation | From start of treatment to post-treatment surveillance scans, up to 6 months
  The Functional Assessment of Cancer Therapy - Head & Neck (FACT-HN) will be used to evaluate quality of life measures at baseline and during treatment. This scale has the sub-categories of physical well being, social/family well-being, emotional well-being, functional well-being, and additional concerns. Each question is scaled from 0 (worst) to 4 (best). Each sub-category will be totaled and a total FACT-HN score will be calculated for each time point. Average sub-category and total scores will be calculated as well as change from baseline to worst scores during treatment.
Total concurrent opioid use using patient reported diaries | From start of treatment to post-treatment surveillance scans, up to 6 months
  Patients will document every dose of opioid medications taken during the study period. This will be used to used to calculated total opioid amounts taken (as oxycodone equivalents) as well as total duration of opioid use in days.
Progression free survival (PFS) | Screening, 3 and 6 month follow up visits
  Progression free survival will be calculated as time to disease progression from start of treatment measured in weeks. This will be documented by PET/CT and/or CT neck and chest completed prior to start of treatment and approximately 3 and 6 months after treatment discontinuation
Overall survival (OS) | From start of treatment up to 18 months
  OS will be calculated as time from start of treatment to death as measured in weeks. This will be documented by survival follow-up during study visits

CONTACTS AND LOCATIONS:
Overall Officials: Jessica McDermott, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No